CLINICAL TRIAL: NCT02420028
Title: A Randomized Controlled Open Label Trial to Assess the Safety and Efficacy of the OptiVein IV Catheter in an Oncologic Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit patients sufficiently
Sponsor: Optomeditech Oy (Industry)
Collaborators: CardioMed Device Consultants, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OMT-CT-003-ONC
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Intravenous Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OptiVein IV catheter (Experimental): Insertion of an IV catheter into the patient's vein, defined as placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.
  Interventions: Device: Insertion of OptiVein IV catheter
- Vasofix Certo IV catheter (Active Comparator): Insertion of an IV catheter into the patient's vein, defined as placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.
  Interventions: Device: Insertion of Vasofix Certo IV catheter

INTERVENTIONS:
Device: Insertion of OptiVein IV catheter — Placement of OptiVein IV catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.
  Arms: OptiVein IV catheter
Device: Insertion of Vasofix Certo IV catheter — Placement of Vasofix Certo IV catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.
  Arms: Vasofix Certo IV catheter

SUMMARY:
A prospective, single-center, open-label, randomized controlled trial to assess the safety and efficacy of the OptiVein IV Catheter in an oncology population. The study hypothesis is that OptiVein IV Catheter use will be superior to the control in successful venous access after first attempt.

DETAILED DESCRIPTION:
The OptiVein IV Catheter is a sterile single use disposable intravascular cannulation device that is modified from CE certified Vasofix Certo Catheter from B.Braun with the additional features of an optical fiber and modified flashplug. The OptiVein System also includes an electronic unit.

The study control and predicate device is the Vasofix Certo IV Catheter from B. Braun Medical Inc. This device is the base device for the OptiVein IV Catheter to which is added the optical fiber and electronic unit.

The OptiVein Catheter shares a similar intended use and the same catheter components as the Vasofix Certo IV Catheter. Clinical data will be obtained to assess if there is a change to the safety and efficacy profile due to the laser component of the OptiVein IV Catheter.

Subject population consists of Oncologic patients who have either difficult to access veins or who have experienced an unsuccessful IV start during their previous visit to the hospital, requiring short-term use of an IV catheter to administer chemotherapy medications intravenously. Subjects may be enrolled multiple times, with each patient-visit being the unit of analysis.

Primary efficacy endpoint is successful IV insertion on the first attempt, defined as placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.

167 and 167 patient-visits will be included in OptiVein or Vasofix Certo respectively (1:1 randomization), resulting in a total sample size of 334 visits. This sample size will provide 80% power to demonstrate the superiority of the OptiVein Catheter to the Vasifix Certo Catheter.

Secondary endpoints include:

1. Total number of attempts required for successful IV insertion.
2. Time to successful IV insertion, defined as time from the first skin puncture to placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal
3. Incidence of blood extravasation resulting in a hematoma
4. Incidence of fluid extravasation delivered through catheter
5. Incidence of infection (phlebitis, dermatitis and induration) at insertion site through 72 hours or at the time of catheter removal, whichever occurs first.
6. Unplanned withdrawal of IV catheter
7. Overall complication rate composed from #3-6 above

ELIGIBILITY:
Inclusion Criteria:

1. Patients on an ongoing chemotherapy program thru peripheral veins delivery
2. Has difficult to access veins (class II or III) OR has experienced an unsuccessful IV start during his/her previous visit to the hospital
3. Requires peripheral IV therapy (catheter)
4. Has an insertion site in the forearm or hand free of deformities, phlebitis, infiltration, dermatitis, burns, lesions or tattoos
5. Demonstrates cooperation with a catheter insertion and the study protocol
6. Patients 18 years of age or greater

Exclusion Criteria:

1. Patients receiving pre-warming of the insertion site
2. Is anesthetized
3. Has a life expectancy of less than one month
4. Transferred from the operating room less than 8 hours post-anasthesia
5. Any patient the research staff deem unobservable
6. The study IV site needs to be immobilized with a splint or other devices
7. Will require a power injection for a radiologic procedure during participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-04-02; Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Successful IV insertion on the first attempt | Immediate
  Successful placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal.

SECONDARY OUTCOMES:
Total number of attempts required for successful IV insertion | Immediate
Time to successful IV insertion | Immediate
  Defined as time from the first skin puncture to placement of the catheter inside the vein allowing for fluid or drug delivery or blood withdrawal
Incidence of blood extravasation resulting in a hematoma | Immediate
Incidence of fluid extravasation delivered through catheter | Immediate
Incidence of infection | After 72 hours or release from hospital, whichever occurs first.
  phlebitis, dermatitis and induration at insertion site through 72 hours or at the time of catheter removal, whichever occurs first.
Unplanned withdrawal of IV catheter | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Tomi Wiklund, M.D, Ph.D., Principal Investigator — Docrates Cancer Center
Locations (1):
- Docrates Cancer Center, Helsinki, Finland